CLINICAL TRIAL: NCT02841930
Title: ActionHealthNYC: A Health Care Access Program for the Uninsured
Brief Title: ActionHealthNYC Research Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: New York City Department of Health and Mental Hygiene (Other Government)
Collaborators: American Institutes for Research (Other); Public Health Solutions (Other); The New York Academy of Medicine (Other); New York City Health and Hospitals Corporation (Other); New York City Human Resources Administration (Unknown); New York City Mayor's Office of Immigrant Affairs (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NYCDOHMH IRB 16-020
Record Dates: First submitted 2016-07-19; First posted 2016-07-22 (Estimated); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Health Services Accessibility
Keywords: Healthcare Access; Undocumented Immigrants; Primary Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Member (Experimental): The member group will be able to join ActionHealth NYC program, where they are assigned a primary care physician and have a standardized fee scale for services obtained in network. Laboratory, diagnostic, and specialty services can be obtained at network H+H locations. They will be offered recommended USPSTF A+B tests/screenings, HIV and TB screening (if indicated), and care coordination. If they are deemed "high risk," enhanced care coordination services will be offered.
  Interventions: Other: ActionHealth NYC
- Study (No Intervention): The study group will be counseled on their options to access health care, including at public hospitals and community health centers. They will receive no additional services from the study.

INTERVENTIONS:
Other: ActionHealth NYC — care coordination, covered preventive services, and standardized costs for ambulatory care
  Arms: Member

SUMMARY:
The ActionHealthNYC program is a year-long demonstration program to improve access to high quality health care for NYC resident immigrants who do not qualify for public insurance with incomes at or below 200% of the Federal Poverty Level (FPL). The purpose of this study is to determine whether improved access and care coordination services provided through the ActionHealth NYC program allows participants to have easier access to healthcare (particularly primary care and preventive services) than non-participants.

DETAILED DESCRIPTION:
The ActionHealthNYC program is a year-long demonstration program to improve access to high quality health care for NYC resident immigrants who do not qualify for public insurance with incomes at or below 200% of the Federal Poverty Level (FPL). Our goal in piloting the program and conducting the research study is to understand the following questions:

* For clients participating in the ActionHealthNYC program, do they report having easier access to health care?
* What are the differences in health care utilization for participants in the ActionHealthNYC program and those not in the program?
* Do the participants in the ActionHealthNYC program report fewer barriers to needed care when compared to those not in the program?
* Are the participants in the ActionHealthNYC program more likely to have received preventive services according to the United States Preventive Services Task Force (USPTF) or recommended services for those with a qualifying condition through their medical home?
* How does the likelihood of receiving a new diagnosis compare between the ActionHealthNYC member group and the study group?
* How does emergency department and hospital use compare between the ActionHealthNYC member group and the study group?

We will be conducting a randomized controlled trial (RCT) where we will be enrolling 2,400 people that meet the eligibility criteria and randomizing half into the ActionHealth NYC program. We will be employing a mixed methods approach to address differences between participants randomized to receive enhanced services through ActionHealthNYC (AHNYC) and those receiving usual care, utilizing surveys, secondary data analysis, key informant interviews and participant focus groups.

ELIGIBILITY:
Inclusion Criteria:

* New York City residents who are uninsured, 19 and older and
* Not currently eligible for Medicaid, Essential Plan, or
* Not currently eligible for private insurance via federal insurance marketplace subsidies due to their immigration status.

Exclusion Criteria:

* Not a New York City resident
* Currently eligible for Medicaid, Essential Plan or private insurance at state exchange with federal subsidies
* Income above 200% of the federal poverty level (FPL)

Enrollees are required to have the NYC Municipal identification card (IDNYC). If they do not have the card, however, they can obtain it and come back for enrollment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2428 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Improved access to healthcare | One year
  e.g. fewer delays in getting needed care

SECONDARY OUTCOMES:
Enhanced healthcare utilization | One year
  e.g. emergency department care utilization rate
Reduced barriers to needed care | One year
  e.g. financial barriers
Enhanced utilization of preventive services | One year
  Utilization of USPSTF recommended services through primary care home
Increased number of new diagnoses | One year

CONTACTS AND LOCATIONS:
Overall Officials: Rishi Sood, MPH, Principal Investigator — New York City Department of Health and Mental Hygiene
Locations (1):
- New York City Department of Health and Mental Hygiene, Long Island City, New York, United States

IPD SHARING:
Plan to Share IPD: No